CLINICAL TRIAL: NCT02956876
Title: Equivalence of Monitoring by a Nurse Practitioner for Patients With Digestive Cancer, Requiring Intravenous Chemotherapy Versus a Medical Monitoring
Brief Title: Equivalence of Monitoring by a Nurse Practitioner for Patients With Digestive Cancer
Acronym: INCISIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2015/211/HP
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: ColoRectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse practitioner consultation (Experimental): standard chemotherapy for colorectal cancer
  Interventions: Drug: standard chemotherapy for colorectal cancer; Other: Nurse practitioner consultation
- Standard consultation (Other): standard chemotherapy for colorectal cancer
  Interventions: Drug: standard chemotherapy for colorectal cancer; Other: Medical practitioner consultation

INTERVENTIONS:
Drug: standard chemotherapy for colorectal cancer — standard chemotherapy for colorectal cancer
Other: Nurse practitioner consultation — Nurse practitioner consultation will be done standard chemotherapy for colorectal cancer
  Arms: Nurse practitioner consultation
Other: Medical practitioner consultation — Medical practitioner consultation will be done standard chemotherapy for colorectal cancer.
  Arms: Standard consultation

SUMMARY:
With 42,150 new cases per year, colorectal cancer is the third cause of cancer in France according to the latest report from the Institut national du Cancer (INCa). Second leading cause of cancer death in men, its management is a public health problem. According to projections by WHO, the prevalence of cancers expected to increase 50% by 2050 especially in digestive oncology. These projections can be concluded that the demand for care will continue to be growing.

Medical advances and societal leading to increased life expectancy, have operated a mutation of the cancer disease. Formerly fatal disease, it is now a chronic disease in some cases. These changes are causing new challenges for the health system.

To address this problem, it is asked health professionals to adapt the organization of health care delivery to improve efficiency, in a constrained economic environment. To this end, action 4.1 of the cancer plan includes the creation of clinical nursing profession, a proposal reiterated in article 120 of the French Health System Law. Nursing clinicians will be empowered to ensure, under certain conditions, prescription treatments protocolized of follow-up tests, further treatment and support, as well as the extension or adaptation of specific treatments.

This project is a first step, in France, in thinking around new organizations in the supply of care in oncology.

For patients, strengthening their monitoring during chemotherapy, will better know their tolerance regarding chemotherapy. This optimized management of chemotherapy-induced effects will help reduce the use of emergency care.

The establishment of such a practitioner will free medical time to handle the most complex patients and perform tasks related to research.

For hospital pharmacies this type of organization will optimize their productivity by anticipating orders for chemotherapy pockets.

This project represents an opportunity to demonstrate the added value of advanced practice nurses in France in the health system and particularly in oncology. It also adds value to clinical expertise nurse and register the profession in the research.

The hypothesis is that the quality and safety of care provided by a nurse practitioner are equivalent to those provided by a doctor at follow-up of patients with gastrointestinal cancer, treated with intravenous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Digestive diagnostic of colorectal cancer.
* Treatment with intravenous chemotherapy or treatment with concomitant oral and intravenous chemotherapy.
* Patient beginning a cycle of chemotherapy he had already received chemotherapy sessions or not.
* Patient aged 18 or over.
* Patient with predictable life expectancy greater than 3 months.
* Patient speak and understand the French.
* Patient having read and understood the information letter and signed the consent form.
* For women of childbearing age: effective contraception 3 months before the start of treatment and negative blood pregnancy test

Exclusion Criteria:

* Patient aged over 80.
* Patient aged under 18.
* Prognosis committed within 3 months.
* Pregnant women or breastfeeding.
* Initial clinical assessment quoting fatigue to a higher grade 2 according to the WHO classification before the start of chemotherapy treatment.
* Against indication(s) for chemotherapy.
* Person deprived of liberty by an administrative or judicial decision or person under the protection of a conservator.
* History of disease or psychological or sensory abnormality that may prevent the patient to understand the requirements for participation in the protocol or preventing it from giving informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
Number of side effects of chemotherapy for WHO grade greater than 2 | Day 7

SECONDARY OUTCOMES:
Quality of life of patients by QLQC-30 questionnaire | Day 7
Number of provisional chemotherapy orders | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MICHEL, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided